CLINICAL TRIAL: NCT03131206
Title: A Phase 1/2 Study of Alectinib in RET-rearranged Non-small Cell Lung Cancer or RET-mutated Thyroid Cancer
Brief Title: A Study of Alectinib in RET-rearranged Non-small Cell Lung Cancer or RET-mutated Thyroid Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed due to slow accrual and lack of efficacy.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Awad, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-080
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: ALK-positive Non-small Cell Lung Cancer (NSCLC); RET-positive Non-small Cell Lung Cancer (NSCLC); RET-positive Thyroid Cancer
Keywords: Non-small cell lung cancer; NSCLC; ALK; RET; alectinib; Thyroid cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms | interventions — alectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 RP2D of alectinib (Experimental): The investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have NSCLC, not everyone who participates in this research study will receive the same dose of the study drug. The dosage will depend on the number of participants who have been enrolled in the study and how well the dosage has been tolerated.
  * Alectinib
  * Oral, BID
  * A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  Interventions: Drug: Alectinib
- Cohort A (Experimental): Participants with RET-rearranged NSCLC with no previous history of RET-TKI therapy.
  * Alectinib
  * Oral, BID, participants will receive the RP2D identified during Phase 1.
  * Each treatment cycle will be defined as 28 consecutive days.
  Interventions: Drug: Alectinib
- Cohort B (Experimental): Participants with RET-rearranged NSCLC with previous history of RET-TKI therapy.
  * Alectinib
  * Oral, BID, participants will receive the RP2D identified during Phase 1.
  * Each treatment cycle will be defined as 28 consecutive days.
  Interventions: Drug: Alectinib
- Cohort C (Experimental): Participants with RET-rearranged thyroid cancer
  * Alectinib
  * Oral, BID, participants will receive the RP2D identified during Phase 1.
  * Each treatment cycle will be defined as 28 consecutive days.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — * Oral, BID
  * Phase I: A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  * Phase II: Participants will be treated at the RP2D identified during Phase I. Each treatment cycle will be defined as 28 consecutive days.
  Other Names: Alecensa

SUMMARY:
This research trial is studying a drug called alectinib as a possible treatment for non-small cell lung cancer (NSCLC) with specific genetic alterations known as ALK or RET rearrangements, and thyroid cancer with RET rearrangements.

DETAILED DESCRIPTION:
This is a Phase I/II research study, which means that researchers are testing different doses of the drug alectinib in participants with cancer to evaluate its safety, determine a safe dosage range, and identify side effects.

The FDA (the U.S. Food and Drug Administration) has approved alectinib as a treatment option for NSCLC, but at a different dosage.

There are two parts to this study, Phase 1 and Phase 2. In Phase 1, patients with ALK or RET rearranged NSCLC will receive different doses of alectinib to determine the highest dose that can be administered without severe or unmanageable side effects. This is called the maximum tolerated dose and will be the recommended dose for the next part of the study, Phase 2. A Phase I clinical trial tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

During Phase 2, participants with RET rearranged NSCLC or thyroid cancer will be given the maximum tolerated dose. During both Phase 1 and Phase 2, the investigators will determine the effect alectinib has on the body, and the effect alectinib has on cancer.

Alectinib belongs to a class of drugs known as tyrosine kinase inhibitors, which stop tyrosine kinases from working. Tyrosine kinases are enzymes that are responsible for activating many proteins in the body's cells. The ALK and RET kinases play an important role in the survival and growth of tumor cells and in the ability of tumor cells to spread to different parts of the body. In laboratory studies and in patients, alectinib has been shown to block the ALK and RET kinases. By blocking these kinases and stopping them from working, it is hoped that alectinib may prevent the survival of tumor cells in addition to stopping their growth and ability to spread.

The purpose of this research study is to learn about the effects of the study drug alectinib, and to find the best dose for treating ALK-positive or RET-positive cancers.

ELIGIBILITY:
Inclusion Criteria:

* Tumor Types:

  * Phase 1: Subjects must have a histologically or cytologically confirmed diagnosis of locally advanced (AJCC Stage IIIB) not amenable to curative therapy or metastatic (AJCC Stage IV) NSCLC that carries a RET rearrangement, as determined by fluorescence in situ hybridization (FISH), reverse transcription polymerase chain reaction (RT-PCR), or next generation sequencing (NGS) via a CLIA-certified local diagnostic test (LDT).

    --- OR-
  * Phase 1: Subjects must have a histologically or cytologically confirmed diagnosis of metastatic (AJCC Stage IV) NSCLC that carries an ALK rearrangement with CNS metastases, as determined by FISH, RT-PCR, immunohistochemistry (IHC), or NGS via a CLIA-certified LDT.
  * Phase 2 Cohorts A&B: Subjects must have a histologically or cytologically confirmed diagnosis of locally advanced (AJCC Stage IIIB) not amenable to curative therapy or metastatic (AJCC Stage IV) NSCLC that carries a RET rearrangement, as determined by FISH, RT-PCR, or NGS via a CLIA-certified LDT.
  * Phase 2 Cohort C (thyroid cancer): Subjects must have a histologically or cytologically confirmed diagnosis of metastatic thyroid cancer (Stage IV) that carries either a RET rearrangement or activating RET mutation, as determined by FISH, RT-PCR, or NGS via a CLIA-certified LDT.
* Disease Status Requirements:

  * Phase 1: Subjects with a RET rearrangement must have had disease progression after at least one prior line of systemic therapy. Subjects with an ALK rearrangement may be either treatment naive or may have received prior treatment, and must have CNS disease present at baseline. Subjects cannot have received more than one prior RET TKI (such as, but not limited to, vandetanib, sorafenib, sunitinib, ponatinib, or cabozantinib). Subjects enrolling to the Phase 1 portion of the trial must not have received prior alectinib therapy.
  * Phase 2:

    * Cohort A: RET-positive NSCLC subjects must have received at least one prior line of therapy, but must be RET TKI-naive.
    * Cohort B: RET-positive NSCLC that has previously been treated with one RET TKI. Subjects cannot have received more than one prior RET TKI and must not have received prior alectinib.
    * Cohort C: RET-positive thyroid cancer, must be radioactive iodine refractory.
* Subjects must have at least one measurable target lesion according to RECIST v1.1.
* Subjects enrolling to the phase 1 portion of the trial who have received a prior RET TKI must be able and willing to undergo a pre-treatment fresh tumor biopsy.
* Subjects enrolling to Cohort B or C of the phase 2 portion of the trial who have received a prior RET TKI must be able and willing to undergo a pre-treatment fresh tumor biopsy.
* All subjects must have archival tissue confirmed as available for enrollment. Subjects who are TKI naive who do not have archival tissue may undergo a fresh tumor biopsy in lieu of the archival tissue requirement. The archival tissue requirement may be waived for subjects after discussion with the principal investigator.
* Age ≥ 18 years.
* ECOG performance status ≤2 (See APPENDIX A)
* Subjects must have normal organ and marrow function as defined below:

Adequate hematologic function

* Absolute neutrophil count ≥1,500/mcL
* Platelets ≥100,000/mcL
* Hemoglobin ≥ 9.0 g/dL -- Adequate renal function
* serum creatinine ≤1.5 x institutional ULN

  ---- OR-
* Estimated glomerular filtration rate (eGFR) ≥45 mL/min/1.73 m2 as calculated using the Modification of Diet Renal Disease Equation (See APPENDIX B)

  * Subjects must have recovered from treatment toxicities to ≤ Grade 1 or to their pretreatment levels. Subjects who have developed interstitial lung disease (ILD) must have fully recovered.
  * For all females of childbearing potential, a negative serum pregnancy test must be obtained within 3 days prior to starting study treatment.
  * For women who are not postmenopausal (≥12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 3 months after the last dose of study drug. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal or postovulation methods) and withdrawal are not acceptable methods of contraception. Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices.
  * For men: agreement to remain abstinent or use a contraceptive method that results in a failure rate of < 1% per year during the treatment period and for at least 3 months after the last dose of study drug. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal or postovulation methods) and withdrawal are not acceptable methods of contraception.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Cytotoxic chemotherapy or immunotherapy within 3 weeks of study entry.
* Oral targeted therapy within 5 half-lives (if known) or 3 weeks (if half-life is unknown) of study entry.
* Phase 1: subjects who have received prior alectinib therapy.
* For enrollment to the phase 1 portion of the trial: Administration of any cytochrome P450 (CYP)3A inhibitors or inducers within 14 days prior to the first dose of alectinib and from Cycle 1 Day 1 - Cycle 2 Day 8 of the phase 1 portion of the trial. Following completion of this period, strong/potent cytochrome P450 (CYP)3A inhibitors or inducers are prohibited while on study. Please see APPENDIX C.
* Radiation therapy (except palliative to relieve bone pain) within 2 weeks of study entry. Palliative radiation (≤10 fractions) must have been completed at least 48 hours prior to study entry. Stereotactic or small field brain irradiation must have completed at least 2 weeks prior to study entry. Whole brain radiation must have completed at least 4 weeks prior to study entry.
* Major surgery within 4 weeks of study entry. Minor surgical procedures (e.g., port insertion) are not excluded, but sufficient time should have passed for wound healing (as determined by the treating investigator).
* Subjects who are receiving any other investigational agents.
* Liver disease characterized by:

  -- ALT or AST > 3 × institutional ULN (≥ 5 × ULN for subjects with concurrent liver metastasis) confirmed on two consecutive measurements

  --- OR-
* Absolute impaired excretory function (e.g., hyperbilirubinemia) or synthetic function or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices

  --- OR-
* Impaired excretory function (e.g., hyperbilirubinemia) or synthetic function or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices

  ---OR-
* Acute viral or active autoimmune, alcoholic, or other types of acute hepatitis
* Subjects with symptomatic CNS metastases who are neurologically unstable and/or require an increased dose of steroid to manage CNS symptoms within 1 week prior to the first day of treatment are excluded.

  * Subjects with brain or leptomeningeal metastases that do not meet the above criteria are allowed.
  * Symptomatic disease is allowed as long as symptoms are controlled and stable.
* History of hypersensitivity to any of the additives in the alectinib drug formulation.
* Subjects with symptomatic bradycardia.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women.
* Any GI disorder that may affect absorption of oral medications in the opinion of the treating investigator, such as malabsorption syndrome or major bowel or stomach resection.
* Subjects who are unable to swallow pills.
* Subjects with a history of a second primary malignancy. Exceptions include: subjects with a history of malignancies that were treated curatively and have not recurred within 3 years prior to study entry; resected basal and squamous cell carcinomas of the skin, and completely resected carcinoma in situ of any type.
* NCI-CTCAE v4.03 Grade 3 or higher toxicities due to any prior therapy (excluding alopecia), which have not shown improvement and are strictly considered to interfere with current study medication.
* Known HIV positivity or AIDS-related illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Awad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of California, Irvine, Irvine, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Phase 1 portion of the study includes 3 dose levels that can be explored: Dose Level 1 (starting dose), Dose Level -1, and Dose Level 2. This study enrolled only to Dose Level 1, therefore the baseline and outcome measures presented are for the DL1 participants only.
Groups:
- Phase 1 RP2D of Alectinib: Alectinib will be administered orally twice daily. A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
- Phase 2 Cohort A: Participants with RET-positive NSCLC with no previous history of RET-TKI therapy.
- Phase 2 Cohort B: Participants with RET-positive NSCLC with previous history of RET-TKI therapy.
- Phase 2 Cohort C: Participants with RET-positive thyroid cancer
Period: Dose Level 1 (600mg BID 7d, 900mg BID)
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C
Started | 5 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Level 2 (900mg BID 7d, 1200mg BID)
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 5 patients enrolled contributed demographic data.
Groups:
- Phase 1 RP2D of Alectinib: Dose Level 1 (starting dose)
- Total: Total of all reporting groups
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C | Total
Number analyzed (Participants) | 5 | 0 | 0 | 0 | 5
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 64] |  |  |  | 60 [36 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  |  | 3
  Male | 2 |  |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  | 0
  Not Hispanic or Latino | 4 |  |  |  | 4
  Unknown or Not Reported | 1 |  |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  | 0
  Asian | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
  Black or African American | 0 |  |  |  | 0
  White | 4 |  |  |  | 4
  More than one race | 0 |  |  |  | 0
  Unknown or Not Reported | 1 |  |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 |  |  |  | 5
Mutation status [Number; unit: participants] — RET rearrangement or ALK rearrangement, as determined by a CLIA-certified test
  participants
    RET-rearranged NSCLC | 4 |  |  |  | 4
    ALK-rearranged NSCLC | 1 |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase 1)
Description: The maximally administered dose (MAD) of the study medication will be defined as the dose level where at least two subjects develop toxicities consistent with a DLT definition. In this situation, the dose level immediately below the MAD will be defined as the MTD.
Time Frame: 28 Days
Population: 5 patients were analyzed for the MTD, but the MTD was not reached due to incomplete enrollment (6 patients required to evaluate MTD, per protocol; study closed to enrollment after 5 participants were enrolled). There were no participants analyzed in the Phase 2 portion of the study (Cohorts A, B, and C), hence why those fields are NA.
Measure: Number; unit: mg
Groups:
- Phase 1 RP2D of Alectinib: The investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have NSCLC, not everyone who participates in this research study will receive the same dose of the study drug. The dosage will depend on the number of participants who have been enrolled in the study and how well the dosage has been tolerated.
  * Alectinib
  * Oral, BID
  * A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  Alectinib: -- Oral, BID
  * Phase I: A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  * Phase II: Participants will be treated at the RP2D identified during Phase I. Each treatment cycle will be defined as 28 consecutive days.
- Cohort A: Participants with RET-rearranged NSCLC with no previous history of RET-TKI therapy.
  * Alectinib
  * Oral, BID, participants will receive the RP2D identified during Phase 1.
  * Each treatment cycle will be defined as 28 consecutive days.
  Alectinib: -- Oral, BID
  * Phase I: A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  * Phase II: Participants will be treated at the RP2D identified during Phase I. Each treatment cycle will be defined as 28 consecutive days.
- Cohort B: Participants with RET-rearranged NSCLC with previous history of RET-TKI therapy.
  * Alectinib
  * Oral, BID, participants will receive the RP2D identified during Phase 1.
  * Each treatment cycle will be defined as 28 consecutive days.
  Alectinib: -- Oral, BID
  * Phase I: A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  * Phase II: Participants will be treated at the RP2D identified during Phase I. Each treatment cycle will be defined as 28 consecutive days.
- Cohort C: Participants with RET-rearranged thyroid cancer
  * Alectinib
  * Oral, BID, participants will receive the RP2D identified during Phase 1.
  * Each treatment cycle will be defined as 28 consecutive days.
  Alectinib: -- Oral, BID
  * Phase I: A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  * Phase II: Participants will be treated at the RP2D identified during Phase I. Each treatment cycle will be defined as 28 consecutive days.
Arm/Group | Phase 1 RP2D of Alectinib | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 5 | 0 | 0 | 0
mg | NA — MTD could not be evaluated as only 5 subjects were enrolled; per protocol, 6 subjects are required to evaluate MTD. |  |  |

2. Primary Outcome: Objective Response Rate
Description: Preliminary evaluation of objective response rate (ORR) of alectinib was assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Per RECIST v1.1 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 8 weeks
Population: Five participants were enrolled to the Phase 1 portion of the study and had imaging assessments performed; these 5 participants were evaluable for response rate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 RP2D of Alectinib | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 5 | 0 | 0 | 0
percentage of participants | 20 [0.52 to 71.63] |  |  |

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Alectinib
Description: AUC pharmacokinetic parameters will be estimated using non-compartmental models. Comparisons across dose levels will be made to assess proportionality.
  Results are incomplete because study closed to accrual early.
Time Frame: 4 months
Population: Data not collected. Trial terminated early due to slow accrual.
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Progression Free Survival
Description: Progression evaluated using RECIST 1.1 Criteria. Results are incomplete because study closed to accrual early.
Time Frame: 2 Years
Population: Data not collected. Trial terminated early due to slow accrual.
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is recorded from start of enrollment through study completion.
Time Frame: OS was calculated at the time of analysis, which was approximately 22 months after the study opened to enrollment.
Population: Number of participants alive at time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 RP2D of Alectinib | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 5 | 0 | 0 | 0
Participants | 1 |  |  |

6. Secondary Outcome: Duration of Response
Description: Response evaluated using RECIST 1.1 Criteria. Results are incomplete because study closed to accrual early.
Time Frame: 2 Years
Population: Data not collected. Trial terminated early due to slow accrual.
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Peak Plasma Concentration (Cmax) of Alectinib
Description: Cmax pharmacokinetic parameters will be estimated using non-compartmental models. Comparisons across dose levels will be made to assess proportionality. Results are incomplete because study closed to accrual early.
Time Frame: 4 months
Population: Data not collected. Trial terminated early due to slow accrual.
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all participants from first dose through the follow-up period. AE data was collected for approximately 22 months on this study.
Description: AE data is available for the 5 patients enrolled to the Phase I portion of the study. Since the study closed early, no participants were enrolled to Phase 2 Cohorts A, B, or C, and AE and mortality data are not available.
Groups:
- Phase 1 RP2D of Alectinib: The investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have NSCLC, not everyone who participates in this research study will receive the same dose of the study drug. The dosage will depend on the number of participants who have been enrolled in the study and how well the dosage has been tolerated. A 7-day lead-in dosing period will be administered at the start of each dose level. Each treatment cycle will be defined as 28 consecutive days.
  The AE data presented here includes all 5 participants which were enrolled to the Phase 1 portion of the study, to Dose Level 1.
- Phase 2 Cohort A: Participants with RET-positive NSCLC with no previous history of RET-TKI therapy. No participants were enrolled to Cohort A.
- Phase 2 Cohort B: Participants with RET-positive NSCLC with previous history of RET-TKI therapy. No participants were enrolled to Cohort B.
- Phase 2 Cohort C: Participants with RET-positive thyroid cancer. No participants were enrolled to Cohort C.
Arm/Group | Phase 1 RP2D of Alectinib | Phase 2 Cohort A | Phase 2 Cohort B | Phase 2 Cohort C
All-Cause Mortality (participants affected / at risk) | 4/5 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 RP2D of Alectinib (N=5) | Phase 2 Cohort A (N=0) | Phase 2 Cohort B (N=0) | Phase 2 Cohort C (N=0)
Anemia (Blood and lymphatic system disorders) | 2 (7) | NA | NA | NA
Chest pain - cardiac (Cardiac disorders) | 1 (1) | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 1 (1) | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 1 (1) | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 (1) | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA | NA | NA
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (2) | NA | NA | NA
Nausea (Gastrointestinal disorders) | 1 (1) | NA | NA | NA
Stomach pain (Gastrointestinal disorders) | 1 (1) | NA | NA | NA
Edema limbs (General disorders) | 1 (3) | NA | NA | NA
Fatigue (General disorders) | 3 (3) | NA | NA | NA
Pain (General disorders) | 2 (3) | NA | NA | NA
Alkaline phosphatase increased (Investigations) | 2 (3) | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 (3) | NA | NA | NA
CPK increased (Investigations) | 1 (4) | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 (1) | NA | NA | NA
Weight loss (Investigations) | 1 (1) | NA | NA | NA
Anorexia (Metabolism and nutrition disorders) | 2 (2) | NA | NA | NA
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | NA | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | NA | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA | NA
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (3) | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | NA | NA | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA | NA
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA | NA
Concentration impairment (Nervous system disorders) | 2 (2) | NA | NA | NA
Headache (Nervous system disorders) | 1 (1) | NA | NA | NA
Lethargy (Nervous system disorders) | 1 (1) | NA | NA | NA
Memory impairment (Nervous system disorders) | 1 (1) | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 (2) | NA | NA | NA
Confusion (Psychiatric disorders) | 2 (2) | NA | NA | NA
Delirium (Psychiatric disorders) | 1 (1) | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 (1) | NA | NA | NA
Hematuria (Renal and urinary disorders) | 1 (2) | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | NA | NA | NA
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT03131206/Prot_SAP_000.pdf